CLINICAL TRIAL: NCT01836276
Title: Understanding Disparities in Quitting in African American and White Smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nikki Nollen, PhD, MA (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Nikki Nollen, PhD, MA, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12990; 1R01DA031815-01A1 (NIH)
Record Dates: First submitted 2013-04-16; First posted 2013-04-19 (Estimated); Results first posted 2018-09-21 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-09

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- African American (AA) Smokers (Experimental): AA smokers received 12 weeks of Varenicline and 6 smoking cessation counseling sessions.
  Interventions: Drug: Varenicline
- White Smokers (Active Comparator): White smokers received 12 weeks of Varenicline and 6 smoking cessation counseling sessions.
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — 1 mg of varenicline twice daily after titration to full strength in the first week following standard dosing guidelines
  Other Names: Chantix®

SUMMARY:
The purpose of this study is to describe the differences in quitting smoking between African Americans (AA) and White smokers treated with varenicline.

DETAILED DESCRIPTION:
While many studies have evaluated the use of drugs for quitting smoking among Whites, few have assessed efficacy with AAs. Racial/ethical differences in smoking are well documented. AAs smoke less than White smokers but experience disproportionately greater smoking disease and death.

Past studies by the researchers in this study looked at how effective other smoking cessation methods are in AAs. These methods included nicotine gum, nicotine patch and buproprion sustained release. This study will be evaluating varenicline in both AA and White smokers. There has not been a study conducted yet to prospectively research AA-White differences in smoking cessation and also to examine potential causal pathways explaining AA-White differences in quitting.

ELIGIBILITY:
Inclusion Criteria:

* Non-Hispanic African American or non-Hispanic White
* ≥ 18 years of age
* Smoked 3-20 cigarettes per day
* Smoked on >25 days of the past 30 days
* Functioning telephone
* Interested in quitting smoking
* Interested in taking 3 months of varenicline
* Willing to complete all study visits

Exclusion Criteria:

* Renal impairment
* Evidence or history of clinically significant allergic reactions to varenicline
* A cardiovascular event in the past month Hospitalization in the past 2 months for any cardiovascular disease, including but not limited to:

  * Angina
  * Myocardial infarction
  * Peripheral vascular disease
  * Stroke
* New onset of chest pain or arrhythmia in the past 2 months
* History of alcohol or drug dependency in the past year
* Major depressive disorder in the last year requiring treatment
* History of panic disorder, psychosis, bipolar disorder, or eating disorders
* Use of tobacco products other than cigarettes in past 30 days
* Use of pharmacotherapy in the month prior to enrollment, including prior use of varenicline
* Pregnant, contemplating getting pregnant, or breastfeeding
* Plans to move from Kansas City during the treatment and follow-up phase
* Another household member enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikki Nollen, PhD, MA, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Swope Health Central, Kansas City, Missouri

REFERENCES:
- [Derived] Chenoweth MJ, Kim YJ, Nollen NL, Hawk LW Jr, Mahoney MC, Lerman C, Knight J, Tyndale RF. Genetic Prediction of Smoking Cessation Medication Side Effects: A Genome-Wide Investigation of Abnormal Dreams on Varenicline. Clin Pharmacol Ther. 2024 Jun;115(6):1277-1281. doi: 10.1002/cpt.3210. Epub 2024 Feb 19. PMID 38369951
- [Derived] Nollen NL, Mayo MS, Saint Onge JM, Scheuermann TS, Cox LS, Chae D, Leavens E, Ahluwalia JS. The effect of area-level disadvantage and race on smoking abstinence in a clinical trial. Exp Clin Psychopharmacol. 2022 Jun;30(3):279-286. doi: 10.1037/pha0000493. Epub 2021 Aug 9. PMID 34370500
- [Derived] El-Boraie A, Chenoweth MJ, Pouget JG, Benowitz NL, Fukunaga K, Mushiroda T, Kubo M, Nollen NL, Sanderson Cox L, Lerman C, Knight J, Tyndale RF. Transferability of Ancestry-Specific and Cross-Ancestry CYP2A6 Activity Genetic Risk Scores in African and European Populations. Clin Pharmacol Ther. 2021 Oct;110(4):975-985. doi: 10.1002/cpt.2135. Epub 2021 Jan 1. PMID 33300144
- [Derived] Peng AR, Swardfager W, Benowitz NL, Ahluwalia JS, Lerman C, Nollen NL, Tyndale RF. Impact of early nausea on varenicline adherence and smoking cessation. Addiction. 2020 Jan;115(1):134-144. doi: 10.1111/add.14810. Epub 2019 Nov 5. PMID 31502736
- [Derived] Nollen NL, Mayo MS, Sanderson Cox L, Benowitz NL, Tyndale RF, Ellerbeck EF, Scheuermann TS, Ahluwalia JS. Factors That Explain Differences in Abstinence Between Black and White Smokers: A Prospective Intervention Study. J Natl Cancer Inst. 2019 Oct 1;111(10):1078-1087. doi: 10.1093/jnci/djz001. PMID 30657926
- [Derived] Nollen NL, Cox LS, Yu Q, Ellerbeck EF, Scheuermann TS, Benowitz NL, Tyndale RF, Mayo MS, Ahluwalia JS. A clinical trial to examine disparities in quitting between African-American and White adult smokers: Design, accrual, and baseline characteristics. Contemp Clin Trials. 2016 Mar;47:12-21. doi: 10.1016/j.cct.2015.12.001. Epub 2015 Dec 5. PMID 26667382

RESULTS

PARTICIPANT FLOW:
Groups:
- African American Smokers: African Americans smokers received 12 weeks of Varenicline and 6 smoking cessation counseling sessions.
  Varenicline: 1 mg of varenicline twice daily after titration to full strength in the first week following standard dosing guidelines
Period: Overall Study
Arm/Group | African American Smokers | White Smokers
Started | 224 | 225
Week 4 | 198 | 186
Week 12 | 183 | 165
Completed | 196 | 174
Not Completed | 28 | 51
Not completed — Lost to Follow-up | 28 | 51

BASELINE CHARACTERISTICS:
Groups:
- African American; White: 12 weeks of varenicline and 6 counseling sessions.
- Total: Total of all reporting groups
Arm/Group | African American | White | Total
Number analyzed (Participants) | 224 | 225 | 449
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (12) | 40.5 (11.2) | 41.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 112 | 224
  Male | 112 | 113 | 225
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 224 | 0 | 224
  White | 0 | 225 | 225
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Cohabitation Status [Count of Participants; unit: Participants]
  Living alone | 142 | 115 | 257
  Living with a partner | 82 | 110 | 192
Employment Status [Count of Participants; unit: Participants]
  Employed full-time | 77 | 142 | 219
  Employed part-time | 41 | 29 | 70
  Not currently employed | 75 | 28 | 103
  Retired | 11 | 5 | 16
  Student/homemaker | 20 | 21 | 41
Education level [Count of Participants; unit: Participants]
  Less than high school (HS) graduate | 30 | 14 | 44
  HS graduate or HS equivalent (GED) | 64 | 44 | 108
  Some college or tech school | 90 | 116 | 206
  College graduate or higher | 40 | 51 | 91
Health insurance that pays for most medical care [Count of Participants; unit: Participants]
  No | 107 | 102 | 209
  Yes | 117 | 123 | 240
Income [Mean (Standard Deviation); unit: Dollars] | 21,293 (15,501) | 35,806 (21,035) | 28,566 (19,840)
Number of people living in house, including self [Mean (Standard Deviation); unit: Cohabitants] | 2.7 (1.6) | 3.0 (1.8) | 2.8 (1.7)
Housing [Count of Participants; unit: Participants]
  Own a home | 38 | 77 | 115
  Rent or stay with others | 186 | 148 | 334
Perceived Health [Count of Participants; unit: Participants]
  Good, fair, or poor | 125 | 113 | 238
  Very good/excellent | 99 | 112 | 211
Percent Federal Poverty Level [Count of Participants; unit: Participants] — % Federal Poverty Level is based on the Department of Health and Human Services Guidelines, published each year in the Federal Register (HHS). It is a calculation of household size (i.e., number of individuals residing in the household) and household income. < or = 100% federal poverty level represents the lowest economic status.
  Participants
    < or = 100% | 115 | 43 | 158
    101%-200% | 72 | 87 | 159
    201%-250% | 15 | 25 | 40
    251%-300% | 9 | 27 | 36
    301%-400% | 13 | 43 | 56
Height in inches [Mean (Standard Deviation); unit: inches] | 66.8 (3.7) | 66.8 (3.9) | 66.8 (3.8)
Weight in pounds [Mean (Standard Deviation); unit: pounds] | 195.3 (51.2) | 182.9 (44.1) | 189.1 (48.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.8 (8.1) | 28.9 (7.1) | 29.8 (7.7)
Waist circumference in inches [Mean (Standard Deviation); unit: inches] | 37.6 (6.7) | 36.3 (6.2) | 37.0 (6.4)
Cigarettes per day [Mean (Standard Deviation); unit: Cigarettes] | 12.5 (5.7) | 16.9 (4.6) | 14.7 (5.7)
Age when you started smoking regularly [Mean (Standard Deviation); unit: years] | 18.5 (6.5) | 16.5 (4.8) | 17.5 (5.8)
Menthol smoker [Count of Participants; unit: Participants]
  Non-menthol | 31 | 166 | 197
  Menthol | 193 | 59 | 252
Longest quit attempt in months [Mean (Standard Deviation); unit: months] | 24.8 (70.9) | 25.3 (51.7) | 25.0 (62.0)
Time to first cigarette [Count of Participants; unit: Participants]
  After 30 minutes | 47 | 57 | 104
  Within 30 minutes | 177 | 168 | 345
Number of your five best friends smoke [Mean (Standard Deviation); unit: friends] | 2.9 (1.8) | 2.7 (1.7) | 2.8 (1.8)
Number of smokers in the home(not including self) [Mean (Standard Deviation); unit: cohabitants] | 0.6 (1.0) | 0.6 (0.8) | 0.6 (0.9)
Partner smoking status [Count of Participants; unit: Participants]
  No partner/spouse | 94 | 78 | 172
  Partner/spouse is a non-smoker | 68 | 69 | 137
  Partner/spouse is a smoker | 62 | 78 | 140
Withdrawal [Mean (Standard Deviation); unit: units on a scale] — Minnesota Withdrawal Scale total score. Scores range from 0-32 with higher scores indicating more withdrawal.
  units on a scale | 5.3 (4.3) | 5.2 (3.1) | 5.3 (3.8)
Craving [Mean (Standard Deviation); unit: units on a scale] — Questionnaire of Smoking Urges-Brief, a 4-item measure of craving. Total scores range from 4-28 with higher scores indicating a greater degree of craving.
  units on a scale | 14.1 (7.9) | 15.3 (6.7) | 14.7 (7.3)
Perceived stress [Mean (Standard Deviation); unit: units on a scale] — Perceived Stress Scale, a 4-item measure of stress. Total scores range from 0-16 with higher scores indicating greater stress.
  units on a scale | 4.5 (2.7) | 3.6 (2.3) | 4.1 (2.6)
Depression [Mean (Standard Deviation); unit: units on a scale] — Depressive symptoms were assessed using the Patient Health Questionnaire-9, a depression screener that assesses frequency over the past 2 weeks ('not at all' to 'nearly every day') of each of the DSM-IV criteria for depression. Total scores range from 0-27 with higher scores indicating greater depressive symptomology..
  units on a scale | 2.1 (3.4) | 1.2 (1.8) | 1.7 (2.7)
Anxiety [Mean (Standard Deviation); unit: units on a scale] — The Generalized Anxiety Disorder Questionnaire-7 assessed frequency ('not at all' to 'nearly every day') of symptoms of generalized anxiety disorder (e.g., on edge, uncontrolled worry, restlessness) experienced over the past two weeks. Total scores range from 0-21 with higher scores indicating more anxiety symptoms.
  units on a scale | 3.0 (3.6) | 2.1 (2.7) | 2.5 (3.2)
Financial strain [Mean (Standard Deviation); unit: units on a scale] — An 8-item Financial Strain questionnaire assessed participant's difficulty with respect to affording food, clothing, major items (e.g., car), furniture, leisure activities, and bills and the amount of money left at the end of the month after covering all bills and expenses (some, just enough, or not enough). Total scores ranged from 8-24 with higher scores indicating greater financial strain.
  units on a scale | 15.6 (4.3) | 14.6 (4.1) | 15.1 (4.2)
Perceived discrimination [Mean (Standard Deviation); unit: units on a scale] — The Everyday Discrimination Scale (Short Version) assessed experiences of discrimination across five daily life situations (i.e., treated with less respect, receive poorer service, people act as if you are not smart, people are afraid of you, and feeling harassed/threatened). Total scores are summarized by counting the number of situations encountered (range of 0-5) and the frequency of encounters (range of 0-25).
  units on a scale
    number of situations encountered | 2.7 (1.6) | 2.6 (1.6) | 2.7 (1.6)
    frequency encountered | 6.8 (5.1) | 5.1 (4.1) | 5.9 (4.9)
Race Consciousness [Count of Participants; unit: Participants] — This single item from the Behavioral Risk Factor Surveillance System 'Reactions to Race Module' measures race consciousness by asking participants to identify the frequency with which they think about their race from 'never' to 'constantly.'
  Participants
    Never | 109 | 158 | 267
    Once a year | 25 | 25 | 50
    Once a month | 22 | 18 | 40
    Once a week | 14 | 17 | 31
    At least daily | 54 | 7 | 61
Perceived social status [Mean (Standard Deviation); unit: units on a scale] — Subjective Social Status was measured using the MacArthur Scale of Subjective Social Status.This mea sure presents a 10-rung ladder with instructions to imagine that it represents where people stand in the U.S., with higher rungs representing people who are the best off (most money, education, respected jobs) and lower rungs representing people who are the worst off. Participants are asked to select the rung (1-10) that represents where they stand in life relative to other people in the U.S. Higher scores indicate greater perceived social status.
  units on a scale | 4.8 (1.5) | 5.0 (1.5) | 4.9 (1.5)
Satisfaction with life [Mean (Standard Deviation); unit: units on a scale] — The 5-item Satisfaction with Life Scale was used to assess cognitive appraisal of global life satisfaction (e.g., my life if close to ideal, if I could live life over, I would change almost nothing). Total scores range from 5-35 with higher scores indicating greater life satisfaction.
  units on a scale | 20.1 (6.3) | 23.8 (5.5) | 22.0 (6.2)
Cynicism/distrust of others' intentions [Mean (Standard Deviation); unit: units on a scale] — Measured using the 8-item cynicism/distrust subscale from the Cook-Medley Hostility Scale.The 8-items focus on cynical distrust and disparaging views of others' intentions (e.g., 'Most people are honest mainly through fear of being caught,' 'Most people lie to get ahead') and have demonstrated good psychometric properties in other studies. Total scores range from 0-8 with higher scores indicating greater distrust of others intentions.
  units on a scale | 5.7 (1.6) | 4.8 (1.7) | 5.3 (1.7)
Neuroticism/proneness to psychological stress [Mean (Standard Deviation); unit: units on a scale] — Neuroticism, an indicator of proneness to psychological distress, was assessed with 4-items from the Neuroticism scale of the NEO Five-Factor Inventory.(92) The 4-items focus on the tendency to feel tense/jittery, worried, helpless, and angry and have demonstrated good psychometric properties in previous studies. Total scores range from 0-48 with higher scores indicating greater proneness to psychological distress.
  units on a scale | 12.6 (7.1) | 12.5 (6.3) | 12.5 (6.7)
Social cohesion and trust [Mean (Standard Deviation); unit: units on a scale] — Perceived neighborhood disadvantage was assessed using the 5-item Social Cohesion and Trust questionnaire, which assessed participant's beliefs about their neighbors trustworthiness, shared values, willingness to help, close-knit connections, and ability to get along with each other. Total scores range from 5-25 with higher scores indicating more perceived neighborhood cohesion.
  units on a scale | 16.2 (4.7) | 17.8 (4.5) | 17.0 (4.7)
Neighborhood problems [Mean (Standard Deviation); unit: units on a scale] — Perceived neighborhood disadvantage was assessed using the 10-item Neighborhood Problems questionnaire, which asked participants to identify the degree to which issues such as litter, vandalism, noise, traffic, and safety are problems in their neighborhood. Total scores range from 10-30 with higher scores indicating more neighborhood problems.
  units on a scale | 15.5 (4.7) | 13.5 (3.4) | 14.5 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cotinine-verified 7-day Point Prevalence Smoking Abstinence at Week 26
Description: Defined as having no cigarettes for the previous 7 days at the Week 26 visit. The recommended cut-off of 15ng/ml for salivary cotinine will be used to differentiate smokers from non-smokers.
Time Frame: Change from Baseline to Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | African American (AA) Smokers | White Smokers
Number analyzed (Participants) | 224 | 225
Participants | 32 | 55

ADVERSE EVENTS:
Time Frame: Adverse events were collected between weeks 0-16.
Groups:
- African American; White: Varenicline treatment began at Week 0 and continued through Week 12. Adverse events were monitored through week 16.
Arm/Group | African American | White
All-Cause Mortality (participants affected / at risk) | 0/224 | 1/225
Serious Adverse Events (participants affected / at risk) | 1/224 | 5/225
Other Adverse Events (participants affected / at risk) | 210/224 | 206/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | African American (N=224) | White (N=225)
Fluid on the heart (Cardiac disorders) | 1 (1) | 0 (0)
Depressive episode (Psychiatric disorders) | 0 (0) | 1 (1)
Seizure (Vascular disorders) | 0 (0) | 1 (1)
Heart attack (Cardiac disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Intestinal blockage (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | African American (N=224) | White (N=225)
Hostility, aggression, or other change in behavior not normal for you (Psychiatric disorders) | 13/220 (13) | 13/214 (13)
Fatigue or loss of energy (General disorders) | 18/220 (18) | 21/214 (21)
Nausea (Gastrointestinal disorders) | 34/220 (34) | 43/214 (43)
Trouble Sleeping (General disorders) | 26/220 (26) | 28/214 (28)
Headaches (General disorders) | 20/220 (20) | 17/214 (17)
Abnormal dreams (General disorders) | 29/220 (29) | 9/214 (9)
Gas or flatulence (Gastrointestinal disorders) | 37/220 (37) | 32/214 (32)
Constipation (Gastrointestinal disorders) | 26/220 (26) | 18/214 (18)
Dizziness (General disorders) | 8/220 (8) | 3/214 (3)
Dry mouth (General disorders) | 18/220 (18) | 17/214 (17)
Irritability (Psychiatric disorders) | 24/220 (24) | 27/214 (27)

LIMITATIONS AND CAVEATS:
Findings cannot be generalized to non-US Blacks and Whites and require replication with smokers outside the Midwestern US. Relative efficacy of varenicline versus placebo cannot be determined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT01836276/Prot_SAP_000.pdf